CLINICAL TRIAL: NCT06730867
Title: Piloting Eye Movement Desensitization and Reprocessing (EMDR) in People Living With HIV and Trauma
Brief Title: Piloting Eye Movement Desensitization and Reprocessing (EMDR) Therapy in People Living With HIV and Trauma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Bethany Rhoten, Assistant Professor, Vanderbilt University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 240542
Record Dates: First submitted 2024-11-20; First posted 2024-12-12 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: HIV Infected Individuals
Keywords: HIV; EMDR; trauma
MeSH Terms: conditions — Wounds and Injuries | interventions — Eye Movement Desensitization Reprocessing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- People Living With HIV (PLHIV) (Experimental)
  Interventions: Behavioral: EMDR Therapy Protocol

INTERVENTIONS:
Behavioral: EMDR Therapy Protocol — The intervention involves an eight-week program that details a specific EMDR protocol and questionnaire for people living with HIV. The EMDR sessions occur once a week for eight weeks under the supervision of the investigator.
  Other Names: Eye Movement Desensitization and Reprocessing

SUMMARY:
Eye Movement Desensitization and Reprocessing therapy is a time-limited trauma-response therapy that treats symptoms of stress that result disturbing life experiences. Eye Movement Desensitization and Reprocessing therapy has been used to treat trauma-related symptoms for people living with HIV. People living with HIV tend to experience higher psychiatric morbidity rates of depression, anxiety, and post-traumatic stress symptoms than the general population. However, even with case studies of Eye Movement Desensitization and Reprocessing therapy on people living with HIV, there is no definitive protocol for the clinician as they navigate the therapy. This study aims to assess the feasibility and acceptability of delivering an Eye Movement Desensitization and Reprocessing therapy protocol tailored for people living with HIV and trauma.

20 people living with HIV will be recruited to participate in an eight-week Eye Movement Desensitization and Reprocessing therapy. The therapy will be focused on assessing the viability of an Eye Movement Desensitization and Reprocessing protocol that is specified for people living with HIV.

DETAILED DESCRIPTION:
People living with HIV experience high psychiatric morbidity with rates of depression, anxiety, and post-traumatic stress symptoms two to three times higher than that of the general population. Compared to the general population, people living with HIV also experience a disproportionately high prevalence of trauma. Trauma can lead to development of post-traumatic stress disorder, mood disorders, and substance use disorder, all of which are associated with poor outcomes with regard to HIV care linkage, care retention, medication adherence, and viral suppression. Eye Movement Desensitization and Reprocessing therapy a time-limited psychotherapy approach that enables people to heal from emotional distress that is the result of disturbing life experiences. The theory underlying Eye Movement Desensitization and Reprocessing therapy is the Adaptive Information Processing Model which suggests that traumatic experiences can overwhelm the brain's natural coping mechanisms, leading to emotional distress. While the biological basis of Eye Movement Desensitization and Reprocessing is still being explored, there is evidence to suggest that it works by increasing cerebral hemisphere connectivity through neuronal activation, similar to those of rapid eye movement and short-wave sleep phases. This exhausts working memory which alters the quality of storage of traumatic memories and reduces the intensity of episodic memories and with this, symptoms of post traumatic stress disorder. Eye Movement Desensitization and Reprocessing therapy facilitates the processing of traumatic memories by accessing and reprocessing them through an eight-phase series of structured techniques. During the desensitizing and reprocessing phase sessions, the Eye Movement Desensitization and Reprocessing therapist guides the client through a series of eye movements or other forms of bilateral stimulation while focusing on the traumatic memory, and the client is encouraged to explore any thoughts, emotions, or physical sensations that arise during the process. Through repeated sessions, Eye Movement Desensitization and Reprocessing helps integrate traumatic memories into a more adaptive, organized form.

Eye Movement Desensitization and Reprocessing has been increasingly used beyond treating post traumatic stress disorder in recent years, and studies have shown its effectiveness in treating other psychological disorders. There is preliminary evidence to suggest that Eye Movement Desensitization and Reprocessing can be a beneficial treatment option for depression and anxiety disorders. Eye Movement Desensitization and Reprocessing protocols have been tailored for specific patient populations including oncology, autism, addiction, combat veterans, sexual abuse survivors, and those who have experienced complex trauma. The use of Eye Movement Desensitization and Reprocessing, however, for relieving HIV-related psychological distress in people living with HIV and trauma is novel. HIV-related psychological distress encompasses changes to emotional status, symptom burden, HIV disclosure distress, and HIV-related stigma.23 Piloting an Eye Movement Desensitization and Reprocessing protocol tailored for people living with HIV and trauma is an important first step in realizing the potential for this modality to relieve HIV-related psychological distress.

Rationale and Specific Aims

The purpose of this project is to assess the feasibility and acceptability of delivering an Eye Movement Desensitization and Reprocessing protocol tailored for people living with HIV and trauma. We hypothesize that delivering an Eye Movement Desensitization and Reprocessing protocol tailored for people living with HIV and trauma will be both feasible and acceptable.

We will recruit 20 people living with HIV and trauma living in Tennessee to complete an eight-session Eye Movement Desensitization and Reprocessing protocol. Session 1 will include Eye Movement Desensitization and Reprocessing Phases 1 and 2 (history taking and treatment preparation and planning). At the end of Session 1, participants will select key targets for reprocessing that include HIV-related and adjacent events. During Sessions 2-8, participants will work through each key target using Eye Movement Desensitization and Reprocessing phases 3-8 (session target selection; desensitization and reprocessing; installation of positive cognition; body scan, closing, and reevaluation).

Specific Aim 1: To assess the feasibility of delivering an Eye Movement Desensitization and Reprocessing protocol tailored for people living with HIV who have experienced trauma. Feasibility will be assessed by a) recruitment of people living with HIV and trauma to participate in Eye Movement Desensitization and Reprocessing; b) level of study retention; c) level of engagement of participants with Eye Movement Desensitization and Reprocessing; and d) Eye Movement Desensitization and Reprocessing therapist ability to deliver Eye Movement Desensitization and Reprocessing with sufficient fidelity to the treatment protocol.

Specific Aim 2: To assess the acceptability of delivering an Eye Movement Desensitization and Reprocessing protocol tailored for people living with HIV who have experienced trauma. Acceptability will be assessed by a) program completion rate; b) data collection completion rates, c) intervention evaluation forms, and d) participant reports.

Inclusion/Exclusion Criteria

Description: A convenience sample of adults aged 18 or greater living with HIV who are at least one year post diagnosis who have also experienced trauma according to the Life Events Checklist will be recruited from the Nashville, TN metro area community via: 1) Nashville CARES HIV Clinic; 2) e-advertisements (e.g. ResearchMatch); and 3) IRB-approved study flyers. Importantly, healthcare providers at Nashville CARES will refer clinic patients to the study and will provide a private space for in-person or virtual (computer provided) Eye Movement Desensitization and Reprocessing sessions. Individuals will be excluded from study participation if they have: 1) current suicidal ideation; 2) a diagnosis of schizophrenia; 3) active psychosis; 4) dissociative identity disorder; 5) current severe major depression; or 6) have previously received Eye Movement Desensitization and Reprocessing therapy. Rationale: The Eye Movement Desensitization and Reprocessing protocol used in this study will be targeted to those who have had their HIV diagnosis for at least one year. Other protocols (outside this study) are more appropriate for targeting more recent events (e.g. a new HIV diagnosis). It would not be appropriate to conduct Eye Movement Desensitization and Reprocessing sessions with individuals experiencing the excluded conditions.

Enrollment/Randomization

Participants will be recruited from the Nashville, TN metro area community via: 1) Nashville CARES HIV Clinic; 2) e-advertisements (e.g. ResearchMatch); and 3) IRB-approved study flyers. Potential participants will be provided the opportunity to self-screen without asking them to disclose any information about themselves prior to consent. We will present the individual with a list of inclusion/exclusion criteria and then ask if they would like to proceed with consent, with the understanding that they aren't proceeding if they don't meet the criteria. Individuals who wish to proceed provide informed consent prior to engaging in any study activities. Participants will then complete the Life Events Checklist for the researcher's review. Individuals who have experienced trauma as reflected by checking any event on the Life Events Checklist and still wish to participate will proceed to completing study baseline surveys. As this is a pilot/feasibility study, we are not using a threshold on the Life Events Checklist. If a participant self-reports experiencing any trauma via checking anything on the Life Events Checklist, they are eligible to participate. Privacy will be maintained by speaking to potentially eligible individuals in a private room or via phone, depending on potential participant preference. Study participants will complete baseline assessments and the research staff will schedule the Eye Movement Desensitization and Reprocessing sessions and location (Wesley Place Clinic, Nashville CARES, or virtual) according to participant preference.

Study Procedures

Participants will be recruited from the Nashville, TN metro area community via: 1) Nashville CARES HIV Clinic; 2) e-advertisements (e.g. ResearchMatch); and 3) IRB-approved study flyers. Potential participants will be able to self-screen for the study by reviewing inclusion and exclusion criteria. Potential participants who self-screen in and wish to participate will provide informed consent prior to engaging in any study activities. Once consent has been obtained, participants will complete the Life Events Checklist to assess trauma exposure. Study participants who have been exposed to trauma according to that checklist will then complete baseline assessments and the research staff will schedule the EMDR sessions and location (Wesley Place Clinic, Nashville CARES, or virtual) according to participant preference.

Participant Data Collection includes demographic characteristics and validated instruments previously used in PLHIV:

Trauma Exposure: The Life Events Checklist (LEC-5) is a self-report checklist that assesses exposure to DSM-5 traumatic events.

PTSD Symptom Severity: The PTSD Checklist (PCL-5) is a 20-item questionnaire, assesses PTSD symptom severity based on DSM-5 criteria.

Depression: The Patient Health Questionnaire (PHQ-9) is a 9-item questionnaire assessing presence and severity of depression.

HIV Medication Adherence: The Simplified Medication Adherence Questionnaire (SMAQ) is a 6-item questionnaire evaluating different aspects of patient compliance with treatment: forgetfulness, routine, adverse events, and a quantification of omissions.

Quality of Life: The World Health Organization Quality of Life Brief Version (WHOQOL-BREF) is a 26-item questionnaire addressing four quality of life domains: physical health, psychological health, social relationships, and environment.

Suicide Risk: The Columbia Suicide Severity Risk Scale (C-SSRS) is a six-item questionnaire that assesses the severity and immediacy of suicide risk.

Eye Movement Desensitization and Reprocessing will be delivered to participants according to Shapiro's eight phase dual attention stimuli protocol with phases adapted or expanded to address the needs of people living with HIV. A total of eight weekly 60 minute sessions will be delivered to each study participant. Session 1 will include Eye Movement Desensitization and Reprocessing Phases 1 and 2 (history taking and treatment preparation and planning). At the end of Session 1, participants will select key targets for reprocessing that include HIV-related and adjacent events. During Sessions 2-8, participants will work through each key target using Eye Movement Desensitization and Reprocessing phases 3-8 (assessment and session target selection; desensitization and reprocessing; installation of positive cognition; body scan, closing, and reevaluation). Study participants will have the option to complete Eye Movement Desensitization and Reprocessing sessions either in person (at Wesley Place Clinic or Nashville CARES) or virtually. Both options allow for study participants to maintain privacy during study participation.

Following the eight weekly sessions, participants will complete post-intervention assessment measures as well as a 20-30-minute interview with study staff that will address barriers and facilitators of study participation as well as likes and dislikes of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals that have lived with HIV for over a year.
2. Age 18 or older
3. Have experienced any type of trauma in their lifetime (for example: physical abuse, verbal abuse, physical neglect, emotional neglect, mental illness, substance addiction, imprisonment, witnessing or experiencing violence, natural disasters)

Exclusion Criteria:

1. have current suicidal ideation
2. diagnosis with schizophrenia
3. have active psychosis
4. diagnosed with dissociative identity disorder
5. have current severe major depression
6. have previously received EMDR therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2024-07-29 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Recruitment of PLHIV and trauma to participate in EMDR | 9 months
  Recruitment will be assessed by the rate of enrollment (participants/month).
Study Retention | 10 months
  Retention will be assessed by counting the number of participants who are retained throughout the study.
Engagement | 10 months
  Engagement will be assessed by counting the number of EMDR sessions attended by participants
Intervention Fidelity | 10 months
  Fidelity will be assessed by the EMDR Fidelity Rating Scale

SECONDARY OUTCOMES:
Program Completion | 10 months
  Completion will be assessed by the number of individuals who complete all planned EMDR sessions.
Data Collection Completion | 10 months
  Data collection completion will be assessed by counting the number of assessments that contain missing data.
Intervention Evaluation | 10 months
  The number of participants who rate the intervention as acceptable.

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No